CLINICAL TRIAL: NCT02988960
Title: A Multicenter, Phase 1, Open-Label, Dose-Escalation Study of ABBV-927 and ABBV-181, an Immunotherapy, in Subjects With Advanced Solid Tumors
Brief Title: A Study of ABBV-927 and ABBV-181, an Immunotherapy, in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M15-862; 2016-002219-16 (EudraCT Number)
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Non-small cell lung cancer (NSCLC); Squamous cell carcinoma of the head and neck (SCCHN); Advanced solid tumor; Cancer; Pancreatic adenocarcinoma; Cutaneous melanoma; ABBV-927; ABBV-181; Budigalimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasms; Melanoma | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Escalating Arm 1: ABBV-927 (Experimental): Participants with solid tumors will receive escalating intravenous (IV) doses of ABBV-927.
  Interventions: Drug: ABBV-927
- Escalating Arm 2: ABBV-927 (Experimental): Participants with solid tumors will receive escalating intratumoral (IT) doses of ABBV-927.
  Interventions: Drug: ABBV-927
- Escalating Arm 3: ABBV-927+ABBV-181 (Experimental): Participants with Non-Small Cell Lung Cancer (NSCLC) will receive escalating IV doses of ABBV-927 and IV doses of ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-181
- Escalating Arm 4: ABBV-927+ABBV-181 (Experimental): Participants with Head and Neck Squamous Cell Carcinoma (HNSCC) will receive escalating IT doses of ABBV-927 and IV doses of ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-181
- Escalating Arm 5 (Japan): ABBV-927 (Experimental): Participants with solid tumors will receive escalating intravenous (IV) doses of ABBV-927.
  Interventions: Drug: ABBV-927
- Escalating Arm 6 (Japan): ABBV-927+ABBV-181 (Experimental): Participants with solid tumors will receive escalating IV doses of ABBV-927 and IV doses of ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-181
- Expansion Arm A: ABBV-927 (Experimental): Additional participants with HNSCC or NSCLC will receive intravenous (IV) doses of ABBV-927.
  Interventions: Drug: ABBV-927
- Expansion Arm B: ABBV-927+ABBV-181 (Experimental): Additional participants with HNSCC will receive IT doses of ABBV-927 and IV doses of ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-181
- Expansion Arm C: ABBV-927+ABBV-181 (Experimental): Additional participants with NSCLC will receive IV doses of ABBV-927 and IV doses of ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-181

INTERVENTIONS:
Drug: ABBV-927 — Intravenous
  Arms: Escalating Arm 1: ABBV-927; Escalating Arm 3: ABBV-927+ABBV-181; Escalating Arm 5 (Japan): ABBV-927; Escalating Arm 6 (Japan): ABBV-927+ABBV-181; Expansion Arm A: ABBV-927; Expansion Arm C: ABBV-927+ABBV-181
Drug: ABBV-927 — Intratumoral
  Arms: Escalating Arm 2: ABBV-927; Escalating Arm 4: ABBV-927+ABBV-181; Expansion Arm B: ABBV-927+ABBV-181
Drug: ABBV-181 — Intravenous
  Other Names: Budigalimab
  Arms: Escalating Arm 3: ABBV-927+ABBV-181; Escalating Arm 4: ABBV-927+ABBV-181; Escalating Arm 6 (Japan): ABBV-927+ABBV-181; Expansion Arm B: ABBV-927+ABBV-181; Expansion Arm C: ABBV-927+ABBV-181

SUMMARY:
This is a dose-escalation study designed to evaluate the safety, pharmacokinetics, and pharmacodynamics of ABBV-927, and to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RPTD) for ABBV-927 when administered as monotherapy or as combination therapy with ABBV-181 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Participants have adequate bone marrow, kidney and liver function.
* Participants with a history of chronic heart failure or significant cardiovascular disease must have an echocardiogram or multigated acquisition scan indicating left ventricular ejection fraction greater than or equal to 45% within 28 days prior to the first dose of study drug.
* Participants must have creatinine clearance greater than or equal to 50 mL/min as measured by 24-hour urine or estimated by the Cockcroft-Gault formula.
* Participants must have total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase and alanine aminotransferase less than or equal to 2.5 times ULN.
* Participants in all monotherapy arms must have an advanced solid tumor that has progressed on standard therapies known to provide clinical benefit or the participants are intolerant to such therapies.
* Participants in all combination therapy arms must have recurrent or metastatic HNSCC or NSCLC and previously received platinum-based therapy and progressed either during or after anti-programmed death ligand 1 (PDL1)-based therapy. In addition, participants must have received only one prior immunotherapy.
* The Sponsor may decide to limit the specific tumor types selected or treatment settings for specific arms based on evidence gathered.

Exclusion Criteria:

* Participant must not have an active or prior documented autoimmune disease in the last 2 years.
* Participant must not have current or prior use of immunosuppressive medication within 14 days prior to the first dose (with certain exceptions).
* Participant must not have a history of primary immunodeficiency, bone marrow transplantation, chronic lymphocytic leukemia, solid organ transplantation, previous clinical diagnosis of tuberculosis, inflammatory bowel disease, interstitial lung disease, or immune-mediated pneumonitis.
* Participant must not have a history of clinically significant uncontrolled condition(s) including but not limited to the following: uncontrolled hypertension; symptomatic congestive heart failure; unstable angina pectoris or cardiac arrhythmia including atrial fibrillation.
* Participant must not have a history of coagulopathy or a platelet disorder associated with significant clinical risk of thromboembolic event in the judgement of the investigator, or major thromboembolic event within 6 months prior to the first dose of study treatment.
* Participant must not have a prior grade greater than or equal to 3 immune-mediated neurotoxicity or pneumonitis while receiving immunotherapy.
* Participant must not have a known uncontrolled malignancy of the central nervous system.
* Participants in all combination therapy arms must not have a history of exposure to an immunotherapy experiencing an immune-mediated adverse event that required permanent discontinuation of the immunotherapy.
* Female participants must not be pregnant, breastfeeding or considering becoming pregnant during the study or for at least 3 or 5 months (for monotherapy and combination therapy participants, respectively) after the last dose of study drug.
* Male participants must not be considering fathering a child or donating sperm during the study or for at least 3 or 5 months (for monotherapy and combination therapy participants, respectively) after the last dose of study drug.
* Participant is judged by the investigator to have evidence of hemolysis.
* For Japan only, participants with a history of interstitial lung disease (pneumonitis) or current interstitial lung disease (pneumonitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended Phase 2 dose (RPTD) for ABBV-927 when administered as monotherapy or as combination therapy with ABBV-181 | Up to 8 weeks
  The MTD and the RPTD of ABBV-927 when administered as monotherapy or as combination therapy with ABBV-181 will be determined during the dose escalation phase of the study. Once the RPTD has been determined, the dose expansion portion will begin.
Time to Cmax (Tmax) of ABBV-927 | Up to 12 weeks after participant's first dose
  Time to Cmax (Tmax) of ABBV-927.
Maximum observed serum concentration (Cmax) of ABBV-927 | Up to 12 weeks after participant's first dose
  Maximum observed serum concentration (Cmax) of ABBV-927.
Terminal-Phase Elimination Rate Constant (β) of ABBV-927 | Up to 12 weeks after participant's first dose
  Terminal-phase elimination rate constant (β)of ABBV-927.
Terminal half-life (t1/2) of ABBV-927 | Up to 4 weeks after participant's first dose
  Terminal half-life (t1/2) of ABBV-927.
Area under the serum concentration-time curve (AUCt) of ABBV-927 | Up to 12 weeks after participant's first dose
  Area under the serum concentration-time curve from time zero to the time of last measurable concentration (AUCt) of ABBV-927.
Time to Cmax (Tmax) of ABBV-181 | Up to 12 weeks after participant's first dose
  Time to Cmax (Tmax) of ABBV-181.
Maximum observed serum concentration (Cmax) of ABBV-181 | Up to 12 weeks after participant's first dose
  Maximum observed serum concentration (Cmax) of ABBV-181.
Terminal-Phase Elimination Rate Constant (β) of ABBV-181 | Up to 12 weeks after participant's first dose
  Terminal-phase elimination rate constant (β)of ABBV-181.
Terminal half-life (t1/2) of ABBV-181 | Up to 4 weeks after participant's first dose
  Terminal half-life (t1/2) of ABBV-181.
Area under the serum concentration-time curve (AUCt) of ABBV-181 | Up to 12 weeks after participant's first dose
  Area under the serum concentration-time curve from time zero to the time of last measurable concentration (AUCt) of ABBV-181.
Number of Participants with Adverse Events | Up to 30 days after and up to 24-month of treatment period
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR, defined as the percentage of participants with a confirmed partial, complete response, or stable disease for at least 24 weeks to the treatment) | Up to 30 days after and up to 24-month of treatment period
  CBR defined as the proportion of subjects with a confirmed partial response (PR), complete response (CR), or stable disease for at least 24 weeks to the treatment.
Duration of objective response (DOR) | Up to 30 days after and up to 24-month of treatment period
  DOR is defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Objective response rate (ORR) | Up to 30 days after and up to 24-month of treatment period
  ORR is defined as the proportion of participants with a confirmed partial or complete response to the treatment.
Progression-free survival (PFS) | Up to 30 days after and up to 24-month of treatment period
  PFS time is defined as the time from the first dose of ABBV-927 to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (22):
- United States (7):
  - The Angeles Clinic and Researc /ID# 156324, Los Angeles, California
  - The University of Chicago Medical Center /ID# 155264, Chicago, Illinois
  - Massachusetts General Hospital /ID# 155267, Boston, Massachusetts
  - Carolina BioOncology Institute /ID# 155265, Huntersville, North Carolina
  - Tennessee Oncology-Nashville Centennial /ID# 158654, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center /ID# 155263, Houston, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 155266, Fairfax, Virginia
- Australia (2):
  - Peninsula Oncology Centre /ID# 164372, Frankston, Victoria
  - Austin Health /ID# 171189, Heidelberg, Victoria
- University Health Network_Princess Margaret Cancer Centre /ID# 200819, Toronto, Ontario, Canada
- France (4):
  - Institut Bergonie /ID# 162665, Bordeaux, Gironde
  - Duplicate_Institut Regional du Cancer /ID# 163609, Montpellier, Herault
  - Centre Leon Berard /ID# 162663, Lyon, Rhone
  - Institut Gustave Roussy /ID# 162666, Villejuif, Val-de-Marne
- Japan (2):
  - National Cancer Center Hospital East /ID# 216870, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 217758, Chuo-ku, Tokyo
- South Korea (2):
  - Seoul National University Hospital /ID# 166291, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 166292, Seoul
- Spain (4):
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 200129, Majadahonda, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 200128, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 200127, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 200975, Valencia

IPD SHARING:
Plan to Share IPD: No